CLINICAL TRIAL: NCT00963248
Title: Surveillance of EBV Infection as a Risk Factor for PTLD in Pediatric and Adult Renal Transplant Recipients - a Multicenter Prospective Study
Brief Title: EBV Infection as a Risk Factor for PTLD in Pediatric and Adult Renal Transplant Recipients
Status: Completed | Type: Observational
Sponsor: Klinik für Kinder- und Jugendmedizin (Other)
Responsible Party: Principal Investigator, Dr. med. Britta Hoecker, EBV in pediatric RTx patients, Klinik für Kinder- und Jugendmedizin
Other Study IDs: BToenshoff002
Record Dates: First submitted 2009-08-20; First posted 2009-08-21 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Epstein-Barr Virus Infections
Keywords: EBV; PTLD; RTx; pediatric
MeSH Terms: conditions — Epstein-Barr Virus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — EDTA plasma for EB viral load, serum for differentiated serology and sodium heparine whole-blood for EBV-specific t cells
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Question:

In which stage of an EBV-infection is a selective reduction of immunosuppressive medication reasonable to minimize the risk for PTLD, without putting the transplant recipient at risk of acute rejection episodes due to under immunosuppression?

Aim of study:

Identification of patients at high-risk for PTLD.

DETAILED DESCRIPTION:
PTLD represents a heterogeneous group of abnormal lymphoid proliferations, generally of B-cells, that occur in the setting of ineffective T-cell function because of pharmacological immunosuppression. Because the vast majority of PTLDs are associated with Epstein-Barr virus (EBV) infection, surveillance of EBV infection may have the potential to prevent the development of PTLD by early intervention. However, the cut-off values of "high" EBV viral load remain badly defined due to a lack of prospective studies and assay standardization. The aim of this ongoing multicenter prospective study is the serial detection of primary EBV infection or reactivation in a homogeneous patient population of pediatric renal transplant recipients during the first 2 years posttransplant by the combined analysis of quantitative EBV viral load by a standardized quantitative PCR technique, EBV serology and EBV-specific T-lymphocytes for the identification of high-risk patients.

ELIGIBILITY:
Inclusion Criteria:

* male and female pediatric and adult renal transplant recipients with written informed consent

Exclusion Criteria:

* psychological illness which does not allow patient to understand the study and participate following his own free will
* no written informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: pediatric (< 18 years) and adult (>= 18 years) kidney allograft recipients
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2003-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
EB viral load, serology and EBV-specific T cell in pediatric (and adult) renal transplant recipients with or without clinical symptoms of EBV, PTLD etc. | 9 years

CONTACTS AND LOCATIONS:
Overall Officials: Burkhard Toenshoff, MD, PhD, Principal Investigator — University Children's Hospital of Heidelberg
Locations (1):
- Britta Hoecker, Heidelberg, Germany

REFERENCES:
- [Derived] Hocker B, Fickenscher H, Delecluse HJ, Bohm S, Kusters U, Schnitzler P, Pohl M, John U, Kemper MJ, Fehrenbach H, Wigger M, Holder M, Schroder M, Billing H, Fichtner A, Feneberg R, Sander A, Kopf-Shakib S, Susal C, Tonshoff B. Epidemiology and morbidity of Epstein-Barr virus infection in pediatric renal transplant recipients: a multicenter, prospective study. Clin Infect Dis. 2013 Jan;56(1):84-92. doi: 10.1093/cid/cis823. Epub 2012 Oct 5. PMID 23042966
- [Derived] Hocker B, Bohm S, Fickenscher H, Kusters U, Schnitzler P, Pohl M, John U, Kemper MJ, Fehrenbach H, Wigger M, Holder M, Schroder M, Feneberg R, Kopf-Shakib S, Tonshoff B. (Val-)Ganciclovir prophylaxis reduces Epstein-Barr virus primary infection in pediatric renal transplantation. Transpl Int. 2012 Jul;25(7):723-31. doi: 10.1111/j.1432-2277.2012.01485.x. Epub 2012 Apr 25. PMID 22533698